CLINICAL TRIAL: NCT02535026
Title: Epidemiological, Prospective and Observational Study on the HER2 Status in Breast Invasive Carcinomas Assessed by Immunohistochemistry (IHC) and Silver In-situ Hybridization (SISH) in a Sample of Latin-American Patients
Brief Title: An Observational Study on Human Epidermal Growth Factor Receptor (HER) 2 Status of Breast Invasive Carcinoma in Latin American Participants
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25371
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Breast Cancer Participants: Breast tissue samples from female participants with a breast cancer diagnosis that undergo an anatomopathological examination of surgical specimens and/or core needle biopsies will be considered for analysis in this study.

SUMMARY:
This is a descriptive, prospective, observational and epidemiological study on participants recently diagnosed with breast cancer to evaluate the HER2 status by IHC and SISH procedures.

ELIGIBILITY:
Inclusion Criteria:

- Anatomopathological samples (surgical specimens or when a surgical sample is not possible, a core needle biopsy may be used) from female participants with a histopathological diagnosis of invasive breast cancer

Exclusion Criteria:

* Samples whose residual material in the paraffin block(s) is insufficient for neoplasm representation in the procedures in this study
* Cancer samples that have received previous chemotherapy treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast tissue samples from female participants with a breast cancer diagnosis that undergo an anatomopathological examination of surgical specimens and/or core needle biopsies when surgery is not possible.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Lima, Peru
- Montevideo, Uruguay

RESULTS

PARTICIPANT FLOW:
Groups:
- Breast Cancer (BC) Participants: Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies were considered for analysis in this study.
Period: Overall Study
Arm/Group | Breast Cancer (BC) Participants
Started | 580
Completed | 580
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were included.
Groups:
- Breast Cancer Participants: Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies were considered for analysis in this study.
Arm/Group | Breast Cancer Participants
Number analyzed (Participants) | 580
Age, Continuous [Median (Full Range); unit: years] | 58 [27 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 580
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Epidermal Growth Factor Receptor 2 (HER2) Status in Breast Cancer Specimens Using Immunohistochemistry (IHC) and Silver In-Situ Hybridization (SISH) Procedures
Description: HER2 status of the collected tissue samples was determined based on the results obtained from IHC test and SISH procedure. The IHC test gives a score of 0 to 3 positive (+) that measures the amount of HER2 receptor protein on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+, it's called "HER2 negative (-)." If the score is 2+, it's called "borderline." A score of 3+ is called "HER2 positive." Tissue samples which had the IHC score of 2+ (borderline) were re-tested using SISH procedure for confirmation of the HER2 status. Tissue samples with SISH test results + were considered as HER2+. Tissue samples for which HER2 status was not determined were considered as HER2 equivocal.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples from all participants who were willing to participate in the study.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants
Number analyzed (Participants) | 580
Number analyzed (Tissue samples) | 580
percentage of participants
  HER2 negative | 79.1
  HER2 positive | 19.8
  HER2 equivocal | 1

2. Primary Outcome: Percentage of Participants With Different Phenotypes of Breast Cancer
Description: Breast cancer phenotypes were classified in to a) Luminal A: tissue samples that were estrogen receptor (ER) + and/or progesterone receptor (PR) +, HER2-, and either histologic grade 1 or 2; b) Luminal B: tissue samples that were ER+ and/or PR+ and HER2+ or ER+ and/or PR+ and HER2- and histologic grade 3; c) HER2 enriched: tissue samples that were ER-, PR-, and HER2+; d) Triple negative: tissue samples that were negative for ER, PR, and HER2. Histological grading was done by Nottingham Histologic Score system based on three factors, a) the amount of gland formation (differentiation), b) the nuclear features (pleomorphism) and c) the mitotic activity. Each of these features is scored from 1-3, and then each score is added to give a final total score ranging from 3-9. The final total score is used to determine the grade in the following way: i) Grade 1 tumors have a score of 3-5, ii) Grade 2 tumors have a score of 6-7, and iii) Grade 3 tumors have a score of 8-9.
Time Frame: Baseline up to 30 months
Population: Included all breast cancer tissue samples for which the phenotype could be identified.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants
Number analyzed (Participants) | 574
Number analyzed (Tissue samples) | 574
percentage of participants
  Luminal A | 31.9
  Luminal B | 35
  HER2 Enriched | 12.1
  Triple Negative | 20.9

3. Primary Outcome: Percentage of Participants With Histological Sub-types of Breast Cancer
Description: Histological subtypes of breast cancer included ductal carcinoma, lobular carcinoma, mucinous carcinoma, mixed carcinoma, metaplastic carcinoma, and others.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples from all participants who were willing to participate in the study.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants
Number analyzed (Participants) | 580
Number analyzed (Tissue samples) | 580
percentage of participants
  Ductal carcinoma | 78.3
  Lobular carcinoma | 10.9
  Mucinous carcinoma | 3.6
  Mixed carcinoma | 1.2
  Metaplastic carcinoma | 1.2
  Others | 4.8

4. Primary Outcome: Percentage of Participants With ER Status (Positive or Negative) Across Different Age Groups
Description: Participants were categorized in to following age groups: a) less than (<) 40 years, b) 40-49 years, c) 50-59 years, d) 60-69 years, e) greater than or equal to (≥) 70 years.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples from all participants who were willing to participate in the study.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Groups:
- Breast Cancer Participants (ER-): Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with ER- status were included in this group.
- Breast Cancer Participants (ER+): Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with ER+ status were included in this group.
Arm/Group | Breast Cancer Participants (ER-) | Breast Cancer Participants (ER+)
Number analyzed (Participants) | 203 | 377
Number analyzed (Tissue samples) | 203 | 377
percentage of participants
  <40 years | 9.4 | 6.4
  40-49 years | 19.7 | 21.8
  50-59 years | 30.0 | 24.4
  60-69 years | 22.7 | 24.4
  ≥70 years | 18.2 | 23.1
Statistical Analysis 1: Comparison: Breast Cancer Participants (ER-) vs Breast Cancer Participants (ER+); ER status association with age groups; Test type: Superiority or Other; p = 0.280, Chi-squared

5. Primary Outcome: Percentage of Participants With ER Status (Positive or Negative) Based on Nuclear Grades
Description: Nuclear pleomorphism was observed and graded accordingly. Grade 1: Nuclei small with little increase in size in comparison with normal breast epithelial cells, regular outlines, uniform nuclear chromatin, little variation in size; Grade 2: Cells larger than normal with open vesicular nuclei, visible nucleoli, and moderate variability in both size and shape; Grade 3: Vesicular nuclei, often with prominent nucleoli, exhibiting marked variation in size and shape, occasionally with very large and bizarre forms.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples from all participants who were willing to participate in the study.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants (ER-) | Breast Cancer Participants (ER+)
Number analyzed (Participants) | 203 | 377
Number analyzed (Tissue samples) | 203 | 377
percentage of participants
  Nuclear grade 1 | 0 | 4.8
  Nuclear grade 2 | 30 | 74
  Nuclear grade 3 | 70 | 21.2
Statistical Analysis 1: Comparison: Breast Cancer Participants (ER-) vs Breast Cancer Participants (ER+); ER status association with nuclear grade; Test type: Superiority or Other; p < 0.001, Chi-squared

6. Primary Outcome: Percentage of Participants With ER Status (Positive or Negative) Based on Lymphovascular Invasion
Description: Lymphovascular invasion is entering of breast cancer cells in to the lymph or vascular/blood channels.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples of all participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants (ER-) | Breast Cancer Participants (ER+)
Number analyzed (Participants) | 203 | 376
Number analyzed (Tissue samples) | 203 | 376
percentage of participants
  Present | 69.5 | 60.1
  Absent | 30.5 | 39.9
Statistical Analysis 1: Comparison: Breast Cancer Participants (ER-) vs Breast Cancer Participants (ER+); ER status association with lymphovascular invasion; Test type: Superiority or Other; p = 0.03, Chi-squared

7. Primary Outcome: Percentage of Participants With PR Status (Positive or Negative) Across Different Age Groups
Description: Participants were categorized in to following age groups: a) <40 years, b) 40-49 years, c) 50-59 years, d) 60-69 years, e) ≥70 years.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples from all participants who were willing to participate in the study.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Groups:
- Breast Cancer Participants (PR-): Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with PR- status were included in this group.
- Breast Cancer Participants (PR+): Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with PR+ status were included in this group.
Arm/Group | Breast Cancer Participants (PR-) | Breast Cancer Participants (PR+)
Number analyzed (Participants) | 290 | 290
Number analyzed (Tissue samples) | 290 | 290
percentage of participants
  <40 years | 5.9 | 9.0
  40-49 years | 15.9 | 26.2
  50-59 years | 30.7 | 22.1
  60-69 years | 26.6 | 21.0
  ≥70 years | 21.0 | 21.7
Statistical Analysis 1: Comparison: Breast Cancer Participants (PR-) vs Breast Cancer Participants (PR+); PR status association with age groups; Test type: Superiority or Other; p = 0.004, Chi-squared

8. Primary Outcome: Percentage of Participants With PR Status (Positive or Negative) Based on Nuclear Grades
Description: as for outcome 5
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples from all participants who were willing to participate in the study.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants (PR-) | Breast Cancer Participants (PR+)
Number analyzed (Participants) | 290 | 290
Number analyzed (Tissue samples) | 290 | 290
percentage of participants
  Nuclear grade 1 | 2.1 | 2.1
  Nuclear grade 2 | 44.5 | 72.8
  Nuclear grade 3 | 53.4 | 23.1
Statistical Analysis 1: Comparison: Breast Cancer Participants (PR-) vs Breast Cancer Participants (PR+); PR status association with nuclear grade; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Primary Outcome: Percentage of Participants With PR Status (Positive or Negative) Based on Lymphovascular Invasion
Description: Lymphovascular invasion is entering of breast cancer cells in to the lymph or vascular/blood channels.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples of all participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants (PR-) | Breast Cancer Participants (PR+)
Number analyzed (Participants) | 290 | 289
Number analyzed (Tissue samples) | 290 | 289
percentage of participants
  Present | 67.9 | 58.8
  Absent | 32.1 | 41.2
Statistical Analysis 1: Comparison: Breast Cancer Participants (PR-) vs Breast Cancer Participants (PR+); PR status association with lymphovascular invasion; Test type: Superiority or Other; p = 0.025, ANOVA

10. Primary Outcome: Percentage of Participants With HER2 Status (Positive or Negative) Across Different Age Groups
Description: as for outcome 7
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples of all participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Groups:
- Breast Cancer Participants (HER2-): Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with HER2- status were included in this group.
- Breast Cancer Participants (HER2+): Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with HER2+ status were included in this group.
Arm/Group | Breast Cancer Participants (HER2-) | Breast Cancer Participants (HER2+)
Number analyzed (Participants) | 459 | 115
Number analyzed (Tissue samples) | 459 | 115
percentage of participants
  <40 years | 6.8 | 9.6
  40-49 years | 21.8 | 18.3
  50-59 years | 23.7 | 36.5
  60-69 years | 23.7 | 24.3
  ≥70 years | 24.0 | 11.3
Statistical Analysis 1: Comparison: Breast Cancer Participants (HER2-) vs Breast Cancer Participants (HER2+); HER2 status association with age groups; Test type: Superiority or Other; p = 0.056, ANOVA

11. Primary Outcome: Percentage of Participants With HER2 Status (Positive or Negative) Based on Nuclear Grades
Description: as for outcome 5
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples of all participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants (HER2-) | Breast Cancer Participants (HER2+)
Number analyzed (Participants) | 459 | 115
Number analyzed (Tissue samples) | 459 | 115
percentage of participants
  Nuclear grade 1 | 3.9 | 0
  Nuclear grade 2 | 62.5 | 41.7
  Nuclear grade 3 | 33.6 | 58.3
Statistical Analysis 1: Comparison: Breast Cancer Participants (HER2-) vs Breast Cancer Participants (HER2+); HER2 status association with nuclear grade; Test type: Superiority or Other; p < 0.001, Chi-squared

12. Primary Outcome: Percentage of Participants With HER2 Status (Positive or Negative) Based on Lymphovascular Invasion
Description: Lymphovascular invasion is entering of breast cancer cells in to the lymph or blood/vascular channels.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples of all participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | Breast Cancer Participants (HER2-) | Breast Cancer Participants (HER2+)
Number analyzed (Participants) | 458 | 115
Number analyzed (Tissue samples) | 458 | 115
percentage of participants
  Present | 65.3 | 57.4
  Absent | 34.7 | 42.6
Statistical Analysis 1: Comparison: Breast Cancer Participants (HER2-) vs Breast Cancer Participants (HER2+); Test type: Superiority or Other; p = 0.129, Chi-squared

13. Primary Outcome: Percentage of Participants With Different Phenotypes of Breast Cancer Across Different Age Groups
Description: Breast cancer phenotypes were classified in to a) Luminal A: tissue samples that were ER+ and/or PR+, HER2-, and either histologic grade 1 or 2; b) Luminal B: tissue samples that were ER+ and/or PR+ and HER2+ or ER+ and/or PR+ and HER2- and histologic grade 3; c) HER2 enriched: tissue samples that were ER-, PR-, and HER2+; d) Triple negative: tissue samples that were negative for ER, PR, and HER2. Participants were categorized in to following age groups: a) <40 years, b) 40-49 years, c) 50-59 years, d) 60-69 years, e) ≥70 years.
Time Frame: Baseline up to 30 months
Population: Included all breast cancer tissue samples for which the phenotype was identified.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Groups:
- BC Participants-Luminal A Phenotype: Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with luminal A phenotype were included in this group.
- BC Participants-Luminal B Phenotype: Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with luminal B phenotype were included in this group.
- BC Participants-HER2 Enriched Phenotype: Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with HER2 phenotype were included in this group.
- BC Participants-Triple Negative Phenotype: Breast tissue samples from female participants with a breast cancer diagnosis that underwent an anatomopathological examination of surgical specimens and/or core needle biopsies with triple negative phenotype were included in this group.
Arm/Group | BC Participants-Luminal A Phenotype | BC Participants-Luminal B Phenotype | BC Participants-HER2 Enriched Phenotype | BC Participants-Triple Negative Phenotype
Number analyzed (Participants) | 183 | 201 | 70 | 120
Number analyzed (Tissue samples) | 183 | 201 | 70 | 120
percentage of participants
  <40 years | 3.3 | 10.4 | 10 | 6.7
  40-49 years | 21.9 | 21.9 | 18.6 | 20
  50-59 years | 19.1 | 28.9 | 38.6 | 25.8
  60-69 years | 25.1 | 23.4 | 20 | 25
  ≥70 years | 30.6 | 15.4 | 12.9 | 22.5
Statistical Analysis 1: Comparison: BC Participants-Luminal A Phenotype vs BC Participants-Luminal B Phenotype vs BC Participants-HER2 Enriched Phenotype vs BC Participants-Triple Negative Phenotype; Breast cancer phenotypes association with age groups; Test type: Superiority or Other; p = 0.003, ANOVA

14. Primary Outcome: Percentage of Participants With Different Phenotypes of Breast Cancer Based on Nuclear Grades
Description: Breast cancer phenotypes were classified in to a) Luminal A: tissue samples that were ER+ and/or PR+, HER2-, and either histologic grade 1 or 2; b) Luminal B: tissue samples that were ER+ and/or PR+ and HER2+ or ER+ and/or PR+ and HER2- and histologic grade 3; c) HER2 enriched: tissue samples that were ER-, PR-, and HER2+; d) Triple negative: tissue samples that were negative for ER, PR, and HER2. Nuclear pleomorphism was observed and graded accordingly. Grade 1: Nuclei small with little increase in size in comparison with normal breast epithelial cells, regular outlines, uniform nuclear chromatin, little variation in size; Grade 2: Cells larger than normal with open vesicular nuclei, visible nucleoli, and moderate variability in both size and shape; Grade 3: Vesicular nuclei, often with prominent nucleoli, exhibiting marked variation in size and shape, occasionally with very large and bizarre forms.
Time Frame: Baseline up to 30 months
Population: Included all breast cancer tissue samples for which the phenotype was identified.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | BC Participants-Luminal A Phenotype | BC Participants-Luminal B Phenotype | BC Participants-HER2 Enriched Phenotype | BC Participants-Triple Negative Phenotype
Number analyzed (Participants) | 183 | 201 | 70 | 120
Number analyzed (Tissue samples) | 183 | 201 | 70 | 120
percentage of participants
  Nuclear grade 1 | 5.5 | 4.0 | 0 | 0
  Nuclear grade 2 | 80.9 | 65.2 | 25.7 | 31.7
  Nuclear grade 3 | 13.7 | 30.8 | 74.3 | 68.3
Statistical Analysis 1: Comparison: BC Participants-Luminal A Phenotype vs BC Participants-Luminal B Phenotype vs BC Participants-HER2 Enriched Phenotype vs BC Participants-Triple Negative Phenotype; Breast cancer phenotypes association with nuclear grades; Test type: Superiority or Other; p < 0.001, ANOVA

15. Primary Outcome: Percentage of Participants With Different Phenotypes of Breast Cancer Based on Lymphovascular Invasion
Description: Breast cancer phenotypes were classified in to a) Luminal A: tissue samples that were ER+ and/or PR+, HER2-, and either histologic grade 1 or 2; b) Luminal B: tissue samples that were ER+ and/or PR+ and HER2+ or ER+ and/or PR+ and HER2- and histologic grade 3; c) HER2 enriched: tissue samples that were ER-, PR-, and HER2+; d) Triple negative: tissue samples that were negative for ER, PR, and HER2. Lymphovascular invasion is entering of breast cancer cells in to the lymph or vascular/blood channels.
Time Frame: Baseline up to 30 months
Population: Included breast cancer tissue samples of all participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | BC Participants-Luminal A Phenotype | BC Participants-Luminal B Phenotype | BC Participants-HER2 Enriched Phenotype | BC Participants-Triple Negative Phenotype
Number analyzed (Participants) | 182 | 201 | 70 | 120
Number analyzed (Tissue samples) | 182 | 201 | 70 | 120
percentage of participants
  Present | 67 | 56.7 | 54.3 | 75.8
  Absent | 33 | 43.3 | 45.7 | 24.2
Statistical Analysis 1: Comparison: BC Participants-Luminal A Phenotype vs BC Participants-Luminal B Phenotype vs BC Participants-HER2 Enriched Phenotype vs BC Participants-Triple Negative Phenotype; phenotypes of breast cancer association with lymphovascular invasion; Test type: Superiority or Other; p = 0.001, ANOVA

16. Primary Outcome: Percentage of Participants With Different Phenotypes of Breast Cancer Based on ER Status
Description: Breast cancer phenotypes were classified in to a) Luminal A: tissue samples that were ER+ and/or PR+, HER2-, and either histologic grade 1 or 2; b) Luminal B: tissue samples that were ER+ and/or PR+ and HER2+ or ER+ and/or PR+ and HER2- and histologic grade 3; c) HER2 enriched: tissue samples that were ER-, PR-, and HER2+; d) Triple negative: tissue samples that were negative for ER, PR, and HER2.
Time Frame: Baseline up to 30 months
Population: Included all breast cancer tissue samples for which the phenotype was identified.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | BC Participants-Luminal A Phenotype | BC Participants-Luminal B Phenotype | BC Participants-HER2 Enriched Phenotype | BC Participants-Triple Negative Phenotype
Number analyzed (Participants) | 183 | 201 | 70 | 120
Number analyzed (Tissue samples) | 183 | 201 | 70 | 120
percentage of participants
  ER Status: Positive | 97.8 | 96 | 0 | 0
  ER Status: Negative | 2.2 | 4 | 100 | 100
Statistical Analysis 1: Comparison: BC Participants-Luminal A Phenotype vs BC Participants-Luminal B Phenotype vs BC Participants-HER2 Enriched Phenotype vs BC Participants-Triple Negative Phenotype; phenotypes of breast cancer association with ER status; Test type: Superiority or Other; p < 0.001, ANOVA

17. Primary Outcome: Percentage of Participants With Different Phenotypes of Breast Cancer Based on PR Status
Description: as for outcome 16
Time Frame: Baseline up to 30 months
Population: Included all breast cancer tissue samples for which the phenotype was identified.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | BC Participants-Luminal A Phenotype | BC Participants-Luminal B Phenotype | BC Participants-HER2 Enriched Phenotype | BC Participants-Triple Negative Phenotype
Number analyzed (Participants) | 183 | 201 | 70 | 120
Number analyzed (Tissue samples) | 183 | 201 | 70 | 120
percentage of participants
  PR Status: Positive | 72.1 | 76.6 | 0 | 0
  PR Status: Negative | 27.9 | 23.4 | 100 | 100
Statistical Analysis 1: Comparison: BC Participants-Luminal A Phenotype vs BC Participants-Luminal B Phenotype vs BC Participants-HER2 Enriched Phenotype vs BC Participants-Triple Negative Phenotype; Phenotypes of breast cancer association with PR status; Test type: Superiority or Other; p < 0.001, ANOVA

18. Primary Outcome: Percentage of Participants With Different Phenotypes of Breast Cancer Based on HER2 Status
Description: as for outcome 16
Time Frame: Baseline up to 30 months
Population: Included all breast cancer tissue samples for which the phenotype was identified.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Tissue samples
Arm/Group | BC Participants-Luminal A Phenotype | BC Participants-Luminal B Phenotype | BC Participants-HER2 Enriched Phenotype | BC Participants-Triple Negative Phenotype
Number analyzed (Participants) | 183 | 201 | 70 | 120
Number analyzed (Tissue samples) | 183 | 201 | 70 | 120
percentage of participants
  HER2 Status: Positive | 0 | 22.4 | 100 | 0
  HER2 Status: Negative | 100 | 77.6 | 0 | 100
Statistical Analysis 1: Comparison: BC Participants-Luminal A Phenotype vs BC Participants-Luminal B Phenotype vs BC Participants-HER2 Enriched Phenotype vs BC Participants-Triple Negative Phenotype; phenotypes of breast cancer association with HER2 status; Test type: Superiority or Other; p < 0.001, ANOVA

19. Primary Outcome: Percentage of Participants With Breast Cancer Phenotypes Among Different Hispanic Countries
Description: as for outcome 16
Time Frame: Baseline up to 30 months
Population: Included all breast cancer tissue samples for which the phenotype was identified.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Number of Tissue samples
Arm/Group | BC Participants-Luminal A Phenotype | BC Participants-Luminal B Phenotype | BC Participants-HER2 Enriched Phenotype | BC Participants-Triple Negative Phenotype
Number analyzed (Participants) | 183 | 201 | 70 | 120
Number analyzed (Number of Tissue samples) | 183 | 201 | 70 | 120
percentage of participants | 31.9 | 35.0 | 12.1 | 20.9

ADVERSE EVENTS:
Description: Collection of adverse events data was not applicable as the present study was non-interventional and performed on breast cancer tissue samples obtained from breast cancer participants.
Arm/Group | Breast Cancer Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.